CLINICAL TRIAL: NCT04453254
Title: The Thermogenic and Metabolic Effects of a Whole Food Meal Versus Its Supplemental Equivalent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1302-333
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Food Meal (Active Comparator): A whole meal consisting of 1 cup 2% milk, 1 cup Kashi Go Lean Original cereal, ¼ cup of almonds, ¼ cup of strawberries, and ¼ cup of raspberries.
  Interventions: Other: Whole Food Meal
- Supplement Food Meal (Active Comparator): A supplemental meal equivalent consisting of 1 cup 2% milk, 20 g whey protein, ½ EAS Myoplex bar, and ½ Balance bar.
  Interventions: Other: Supplement Food Meal

INTERVENTIONS:
Other: Whole Food Meal — Isocaloric/ macronutrient whole food meal
  Arms: Whole Food Meal
Other: Supplement Food Meal — Isocaloric/ macronutrient supplement food meal
  Arms: Supplement Food Meal

SUMMARY:
There is limited research on the amount of calories burned and metabolic differences of a complete supplemental meal in comparison to a whole food meal. The purpose of this study is to analyze the differences in calories burned and metabolic response post-consumption of a meal consisting of whole foods compared to its nutritionally engineered equivalent. Investigators hypothesize that energy expenditure and satiety will be greater following consumption of the whole food meal compared to the supplement meal, whereas, there will be no difference in levels of glucose between the two conditions.

DETAILED DESCRIPTION:
Over 50% of U.S. adults today use some form of dietary supplementation to obtain their nutrient intake. Previous research has shown that certain nutritional supplements may produce varying metabolic and thermogenic (calories burned) responses, when compared to other food sources. The difference in thermogenic response may also suggest that there is a difference between a whole food meal and its supplemental equivalent. If there is a difference in thermogenic response, this may indicate that a meal-replacing supplement, such as a ready-to-drink-shake and/or food bar may not induce the same health benefits as a whole food meal in terms of nutrient digestion, absorption, metabolism and storage. There has not been extensive research on the thermic effect and metabolic differences of a complete supplemental meal in comparison to a whole food meal. The purpose of this study is to analyze the differences in thermogenic and metabolic response post-consumption of a meal consisting of whole foods compared to its supplemental, engineered equivalent. It's hypothesized that energy expenditure and satiety will be greater following the whole food meal compared to the supplement meal, whereas, there will be no difference in levels of glucose between the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy females

Exclusion Criteria:

* Participants with specific dietary needs.
* Those with diabetes, impaired fasting glucose, low blood sugar (hypoglycemia) and participants who are classified as high risk.
* Participants with lactose intolerance.
* Participants who regularly use dietary supplements.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
Thermic effect of meals (TEM) also known as postprandial thermogenesis | Baseline line, 15-30, 45-60, 75-90 105-120 minutes postprandial
  The total amount of calories burned after each meal will be measured using indirect calorimetry with the ventilated hood technique. Following meal ingestion, participants will rest quietly for 2 hours during which time their resting energy expenditure will be measured every other 15 minutes for 15 minutes. For example, they will have their resting energy expenditure measured during minutes 15-30, 45-60, 75-90 105-120 following meal ingestion.

SECONDARY OUTCOMES:
Change in blood glucose | Baseline line, 30, 60, 90, 120 minutes postprandial
  Measure the change in postprandial blood glucose compared baseline using the finger stick procedure.
Change in self-reported feelings of hunger, fullness, satiation | Baseline to 120 minutes postprandial
  Visual analog scale of hunger, fullness and satiation using a 100 mm line which subjects place a mark. Closer to 0 mm indicates no feeling at a ll, 100 mm indicates extreme feelings.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acheson KJ, Blondel-Lubrano A, Oguey-Araymon S, Beaumont M, Emady-Azar S, Ammon-Zufferey C, Monnard I, Pinaud S, Nielsen-Moennoz C, Bovetto L. Protein choices targeting thermogenesis and metabolism. Am J Clin Nutr. 2011 Mar;93(3):525-34. doi: 10.3945/ajcn.110.005850. Epub 2011 Jan 12. PMID 21228266
- [Background] Bailey RL, Gahche JJ, Lentino CV, Dwyer JT, Engel JS, Thomas PR, Betz JM, Sempos CT, Picciano MF. Dietary supplement use in the United States, 2003-2006. J Nutr. 2011 Feb;141(2):261-6. doi: 10.3945/jn.110.133025. Epub 2010 Dec 22. PMID 21178089